CLINICAL TRIAL: NCT04140799
Title: Ultrasound Prediction For Vocal Cord Dysfunction In Patients Scheduled For Anterior Cervical Spine Surgeries: A Prospective Cohort Study
Brief Title: Ultrasound Prediction For Vocal Cord Dysfunction In Patients Scheduled For Anterior Cervical Spine Surgeries
Status: Completed | Type: Observational
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Alshaimaa Abdel Fattah Kamel, lecturer of Anaesthesia ,and surgical intensive care, Zagazig University
Other Study IDs: 5645
Record Dates: First submitted 2019-10-16; First posted 2019-10-28 (Actual); Last update posted 2020-06-30 (Actual); Status verified 2020-06

CONDITIONS: Vocal Cord Dysfunction
MeSH Terms: conditions — Vocal Cord Dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: vocal cord ultrasonography — assess vocal cord motion and recurrent nerve function by Transcutaneous laryngeal Ultrasonography in patients scheduled for anterior cervical spine surgeries

SUMMARY:
• Anterior cervical discectomy and fusion (ACDF) is a highly effective and safe method for spinal cord and cervical root decompression. Vocal cord paralysis secondary to recurrent laryngeal nerve injury is a common complication after ACDF. The incidence reported as high as 22%. The standard technique for vocal cord evaluation and the most commonly used tool is direct laryngoscopy. Laryngoscopy causes patients annoyance and could potentially contribute to poor patient compliance. Ultrasonography is a non-invasive technique that is used as an alternative tool.

DETAILED DESCRIPTION:
1. Design: A prospective cohort study.
2. Sample size: Assuming that the target population is 240 and positive predictive value of transcutaneous laryngeal ultrasonography is 89.4%. So, the sample size is 91 cases using OPEN Source Epidemiologic Statistics for Public Health (OPENEPI) with confidence interval 95% and power of test is 80%.

All patients underwent transcutaneous laryngeal ultrasonography examination by both anterior and lateral approach of the Vocal Cords (VCs) before the surgery, immediately after extubation, 2 h, 12h, 24 and 48hour postoperatively by an anesthesiologist with an experience of at least three years in ultrasonography scan.

ELIGIBILITY:
Inclusion Criteria:

* Patient acceptance.
* Both sex
* Age (21-60) years old.
* American Society of Anesthesiologist I / II
* Elective anterior cervical spine surgeries
* patient With Body Mass index (25-35 kg/m²)

Exclusion Criteria:

* Patient refusal.
* Altered mental status.
* Patients with per-existing neurological or thyroid disease affecting vocal cord function.
* Patients with a diagnosis of primary untreated laryngeal/hypopharyngeal cancer.
* Patient with a history of thyroidectomy affecting recurrent laryngeal nerve.
* Patient with a history of laryngeal trauma.
* Pre-operative voice abnormalities.

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Egyptian population scheduled for anterior cervical surgeries
Sampling Method: Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2019-01-16 (Actual); Primary Completion 2020-02-01 (Actual); Study Completion 2020-02-15 (Actual)

PRIMARY OUTCOMES:
Predictive performance associated with the postoperative quantitative trans-cutaneous laryngeal ultrasound: conventional middle approach compared to lateral approach | at the end of the first 48 hours after the surgery
  The predictive performance of postoperative vocal cord edema and paralysis using the conventional middle and lateral approach of trans cutaneous laryngeal ultrasound will be evaluated using sensitivity, specificity and accuracy . the gold standard for diagnosis of vocal cord edema and paralysis will be the rigid laryngoscopy

SECONDARY OUTCOMES:
Diagnostic performance associated with the postoperative quantitative trans-cutaneous laryngeal ultrasound | At 2 weeks and 3 months after the surgery
  The diagnostic performance of postoperative vocal cord paralysis using the trans cutaneous laryngeal ultrasound for diagnosis of recovery of vocal cord paralysis , among subject with vocal cord paralysis
The patient discomfort to procedure | at the end of first 48 hour postoperative
  The patient discomfort to sonography and rigid laryngoscopy by Discomfort score(Visual analogue scale (VAS)) regarding the amount of discomfort experienced during the procedure. Discomfort was reported by placing a mark on a 10-cm line, with the ends representing "not at all uncomfortable" and "extremely uncomfortable."

CONTACTS AND LOCATIONS:
Overall Officials: Alshaimaa A Kamel, M.D, Principal Investigator — Zagazig University
Locations (1):
- Zagazig University, Faculty of medicine, Zagazig, Egypt

REFERENCES:
- [Derived] Kamel AAF, Amin OAI, Hassan MAMM, Elmesallamy WAEA, Hassan EM. Ultrasound prediction for vocal cord dysfunction in patients scheduled for anterior cervical spine surgeries: a prospective cohort study. J Clin Monit Comput. 2021 Aug;35(4):869-875. doi: 10.1007/s10877-020-00546-3. Epub 2020 Jun 15. PMID 32556843